CLINICAL TRIAL: NCT03161379
Title: A Phase II Clinical Trial of GVAX Pancreas Vaccine (With Cyclophosphamide) in Combination With Nivolumab and Stereotactic Body Radiation Therapy (SBRT) Followed by Definitive Resection for Patients With Borderline Resectable Pancreatic Adenocarcinoma
Brief Title: GVAX Pancreas Vaccine (With CY) in Combination With Nivolumab and SBRT for Patients With Borderline Resectable Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1756; IRB00130075 (Other: JHM IRB)
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Cancer
Keywords: Neoadjuvant therapy; immunotherapy; Cytoxan; Cyclophosphamide; Pancreatic Vaccine; SBRT; GVAX; Nivolumab; borderline resectable; Radioimmunotherapy; Vaccine; Antibody; Anti-PD-1
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cyclophosphamide; Nivolumab; Radiosurgery

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CY, Nivolumab, GVAX, and SBRT (Experimental): CY, Nivolumab, GVAX, and SBRT
  Interventions: Drug: Cyclophosphamide; Drug: Nivolumab; Drug: GVAX Pancreas Vaccine; Radiation: Stereotactic Body Radiation (SBRT)

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 200 mg/m2 will be administered one day prior to vaccination (day 0). First dose will be given within 4 to 6 weeks after chemotherapy. 3 weeks after the first dose of immunotherapy the second dose will be given.
  Other Names: CY
Drug: Nivolumab — Nivolumab (240 mg) will be administered one day prior to vaccination. First dose will be given within 4 to 6 weeks after chemotherapy. 3 weeks after the first dose of immunotherapy the second dose will be given.
  Other Names: OPDIVO
Drug: GVAX Pancreas Vaccine — Vaccine will be administered one day after cyclophosphamide and nivolumab. 3 weeks after the first dose of immunotherapy the second dose will be given.
  Other Names: PANC 10.05 pcDNA-1/GM-Neo and PANC 6.03 pcDNA-1/GM-Neo vaccine
Radiation: Stereotactic Body Radiation (SBRT) — SBRT (6.6 Gy over 5 days) will be started during the second dose of immunotherapy (3 weeks after the first dose of immunotherapy).

SUMMARY:
The purpose of this study is to evaluate the safety and clinical activity of FOLFIRINOX along with a whole cell vaccine with immune modulating doses of cyclophosphamide and nivolumab combined with Stereotactic Body Radiation Therapy (SBRT) in patients with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically proven pancreatic cancer that is borderline resectable
* No more than 1 month/cycle (28 days) of systemic therapy for pancreatic cancer
* Age >18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests.
* Woman of child bearing potential must have a negative pregnancy test.
* Must use an acceptable form of birth control while on study.
* Must be candidate for Stereotactic Body Radiation Therapy (SBRT)
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Had major surgery within the last 28 days
* Had an investigational drug or device within the past 28 days
* Prior treatment with immunotherapy agents (including, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4, etc)
* Completed more than 1 month/cycle (28 days) of chemotherapy for pancreas cancer
* Patient on an immunosuppressive systemic treatment, such as steroids, in the past 2 years.
* Other cancer diagnosis requiring treatment within two years
* History of allergic reactions related to the drugs (Nivolumab, Cyclophosphamide, GM-hetastarch, corn, dimethyl sulfoxide, fetal bovine serum, trypsin (porcine origin), yeast or any other component of the GVAX vaccine) in this study.
* Patients receiving growth factors within the last 14 days.
* Currently have or have history of certain study-specified heart, liver, kidney, lung, neurological, psychological, immune or other medical conditions.
* Pregnant or breastfeeding.
* Have known history of infection with HIV, hepatitis B, or hepatitis C.
* Unwilling or unable to follow the study schedule for any reason.
* Presence of tissue or organ allograft, regardless of need for immunosuppression (including corneal allograft)
* Squamous pancreatic cancer or adenosquamous pancreatic cancer with malignant squamous cells >30%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Laheru, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Arsen Osipov, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with borderline resectable pancreatic cancer were enrolled on the study prior to starting standard of care chemotherapy. After completing chemotherapy, participants were re-screened to determine if they were eligible to continue on the study and receive study drug.
Groups:
- CY, Nivolumab, GVAX, and SBRT: Participants received a total of two cycles of Cylophosphamide (CY), Nivolumab, and GVAX Pancreas Vaccine, starting 4-6 weeks after completion of standard of care chemotherapy. Stereotactic Body Radiation Therapy (SBRT) was given over 5 days concurrently with the start of the second cycle. Patients were then evaluated for surgery, and if eligible, had their pancreas tumors resected.
  Cyclophosphamide: 200 mg/m2 IV over 30 minutes on Day 1 of each 21-day cycle.
  Nivolumab: 240 mg IV over 60 minutes on Day 1 of each 21-day cycle.
  GVAX Pancreas Vaccine: 5x10^8 cells, given as 6 intradermal injections (2 on each thigh and 2 on the non-dominant arm), given on Day 2 of each cycle.
  Stereotactic Body Radiation (SBRT): 6.6 Gy over 5 days
Period: Overall Study
Arm/Group | CY, Nivolumab, GVAX, and SBRT
Started (Started = enrolled onto the study) | 31
Completed (Completed = received at least one dose of study drug) | 18
Not Completed | 13
Not completed — Withdrawal by Subject | 4
Not completed — disease progression during chemotherapy | 5
Not completed — no longer surgical candidate after chemotherapy | 2
Not completed — not eligible to start study drug after chemotherapy | 2

BASELINE CHARACTERISTICS:
Arm/Group | CY, Nivolumab, GVAX, and SBRT
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 62 [49 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG scale measures performance status, with scores ranging from 0-5; 0= fully active, performs without restriction, 1= can ambulate, but restricted in physically strenuous activity, 2= ambulatory and capable of self-care, but unable to work, active for >50% of waking hours, 3= limited self-care, confined to bed or chair for >50% of waking hours, 4= completely disabled, totally confined to bed/chair, 5= deceased
  Participants
    ECOG 0 | 16
    ECOG 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: CD8+ T Cell Density in Tumor Tissue
Description: Mean CD8+ T cell density [log(cells per mm^2)], found in resected surgical tissue by Immunohistochemistry (IHC).
Time Frame: evaluated at time of surgery, approximately 2 months from first dose of study drug
Population: Only participants who received study drug, completed surgical resection, and had sufficient tissue to perform IHC analysis. Of the 18 participants treated on study, 13 had sufficient tissue to perform CD8 analysis.
Measure: Mean (Standard Deviation); unit: log (cells per mm^2)
Arm/Group | CY, Nivolumab, GVAX, and SBRT
Number analyzed (Participants) | 13
log (cells per mm^2) | 5.4 (0.8)

2. Secondary Outcome: Pathologic Complete Response (pCR) Rate at Surgical Resection
Description: Number of patients with a pathologic complete response (pCR) rate at surgical resection. A pCR is defined as no viable residual tumor remaining at the time of evaluation.
Time Frame: Assessed at time of surgical resection, approximately 2 months after first dose of study drug
Population: Only participants who received study drug and completed surgical resection are included. Of the 18 participants treated on study, 14 completed surgical resection.
Measure: Count of Participants; unit: Participants
Arm/Group | CY, Nivolumab, GVAX, and SBRT
Number analyzed (Participants) | 14
Participants | 1

ADVERSE EVENTS:
Time Frame: Up to 20 weeks
Description: Adverse events and All Cause Mortality were collected for any patient that received at least one dose of study drug. Of the 31 patients that enrolled, 18 received study drug and were evaluable for adverse events.
Arm/Group | CY, Nivolumab, GVAX, and SBRT
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CY, Nivolumab, GVAX, and SBRT (N=18)
bile duct stenosis (Hepatobiliary disorders) | 1 (1)
sepsis (Infections and infestations) | 1 (1)
skin infection (Infections and infestations) | 1 (1)
weight loss (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CY, Nivolumab, GVAX, and SBRT (N=18)
anemia (Blood and lymphatic system disorders) | 1 (1)
hyperthyroidism (Endocrine disorders) | 1 (1)
hypothyroidism (Endocrine disorders) | 1 (1)
blurred vision (Eye disorders) | 1 (1)
dry eye (Eye disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 5 (6)
bloating (Gastrointestinal disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 3 (5)
dyspepsia (Gastrointestinal disorders) | 1 (1)
flatulence (Gastrointestinal disorders) | 2 (2)
blood in stool (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 4 (7)
upper gastrointestinal hemorrage (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 4 (6)
chills (General disorders) | 1 (1)
edema limbs (General disorders) | 1 (1)
fatigue (General disorders) | 3 (4)
flu-like symptoms (General disorders) | 1 (1)
infusion related reaction (Injury, poisoning and procedural complications) | 2 (2)
pain at site of biopsy (Injury, poisoning and procedural complications) | 1 (1)
alanine aminotransferase increased (Investigations) | 2 (4)
alkaline phosphatase increased (Investigations) | 1 (3)
aspartate aminotransferase increased (Investigations) | 2 (4)
creatinine increased (Investigations) | 1 (1)
hypokalemia (Investigations) | 1 (1)
neutrophil count decreased (Investigations) | 1 (2)
platelet count decreased (Investigations) | 2 (2)
weight loss (Investigations) | 1 (1)
white blood cell decreased (Investigations) | 1 (3)
anorexia (Metabolism and nutrition disorders) | 3 (5)
dehydration (Metabolism and nutrition disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
dizziness (Nervous system disorders) | 2 (2)
headache (Nervous system disorders) | 1 (1)
peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
confusion (Psychiatric disorders) | 1 (1)
breast pain (Reproductive system and breast disorders) | 1 (1)
voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
rash maculopapular (Skin and subcutaneous tissue disorders) | 4 (4)
urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
hot flashes (Vascular disorders) | 1 (1)
hypertension (Vascular disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
vaccine site discoloration (General disorders) | 1 (1)
erythema at vaccine site (General disorders) | 14 (21)
induration at vaccine site (General disorders) | 7 (7)
peeling skin at vaccine site (General disorders) | 1 (1)
pruritus at vaccine site (General disorders) | 12 (17)
swelling at vaccine sites (General disorders) | 5 (11)
tenderness at vaccine site (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT03161379/Prot_SAP_000.pdf